CLINICAL TRIAL: NCT05326620
Title: PROspective Renal Cancer Cohort (PRO-RCC)
Brief Title: National PROspective Infrastructure for Renal Cell Carcinoma (PRO-RCC)
Acronym: PRO-RCC
Status: Recruiting | Type: Observational
Sponsor: PROspective Renal Cancer Cohort Foundation (Other)
Collaborators: Comprehensive Cancer Centre The Netherlands (Other); Merck Sharp & Dohme LLC (Industry); Bristol-Myers Squibb (Industry); Ipsen (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021_218
Record Dates: First submitted 2022-03-17; First posted 2022-04-13 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Renal Cancer; Renal Cell Carcinoma; Renal Cell Cancer Metastatic
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- localized RCC: all patients with localized RCC
- metastatic RCC: all patients with metastatic RCC, synchronous or metachronous

SUMMARY:
PRO-RCC is a nationwide long-term cohort for the collection of real-world clinical data, patient reported outcome measures (PROMs) and patient reported experience measures (PREMs) that provides an infrastructure for observational research and (randomized) interventional studies with the TwiCs (Trial within cohorts) design.

DETAILED DESCRIPTION:
PRO-RCC is designed as a multicenter cohort for all Dutch patients with localized RCC or metastatic renal cell carcinoma (mRCC). The clinical data collection is embedded in the framework of the Netherlands Cancer Registry (NCR). Next to the standardly available data on RCC, additional clinical data will be collected. The informed consent for PRO-RCC covers the online collection of PROMs and PREMS, data sharing and data linking with the NCR. PROMS entail Health-Related Quality of Life (HRQoL), and optional return to work- questionnaires. PREMS entail satisfaction with care. Both PROMS and PREMS are collected through the PROFILES registry and are accessible for the patient and the treating physician. Importantly, participants may also consent to participation in a 'Trial within cohort' studies (TwiC). The TwiC design provides a method to perform (randomized) studies within the registry.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed patients with RCC or synchronous metastatic RCC
* metachronous metastasized RCC
* age >18 years
* capable of understanding Dutch language

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with newly diagnosed (m)RCC can be included, or with synchronous metastasized RCC
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
survival | 5 years
  overall survival
progression | 5 years
  local or distant recurrence
patient reported outcome measures (PROMS) | 5 years
  measured with the EORTC QLQ-C30 questionnaire, every three months in the first year, then yearly up to five years.

SECONDARY OUTCOMES:
Patient reported outcomes of adverse events | 2 years
  Measured with the PRO-CTCAE (patient-reported outcomes version of the common terminology criteria for adverse events), weekly during systemic therapy. Symptoms are scored through 0 (absent) to 3 (severe)

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan Bins, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (26):
- Netherlands (26):
  - Amsterdam UMC locatie VUMC, Amsterdam, North Holland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Meander Medisch Centrum, Amersfoort
  - Gelre ziekenhuis, Apeldoorn
  - Rijnstate, Arnhem
  - Amphia Ziekenhuis, Breda
  - Deventer Ziekenhuis, Deventer
  - Albert Schweitzer, Dordrecht
  - Catharina ziekenhuis, Eindhoven
  - Maxima MC, Eindhoven
  - Treant, Emmen
  - UMCG, Groningen
  - Spaarne Gasthuis, Haarlem
  - Tergooi MC, Hilversum
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Maastricht UMC, Maastricht
  - St Antonius Ziekenhuis, Nieuwegein
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Bravis ziekenhuis, Roosendaal
  - Erasmus MC, Rotterdam
  - Maasstad ziekenhuis, Rotterdam
  - St. Franciscus ziekenhuis, Rotterdam
  - Haaglanden Medisch Centrum, The Hague
  - UMC Utrecht, Utrecht
  - Viecuri, Venray
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yildirim H, Widdershoven CV, Aarts MJ, Bex A, Bloemendal HJ, Bochove-Overgaauw DM, Hamberg P, Herbschleb KH, van der Hulle T, Lagerveld BW, van Oijen MG, Oosting SF, van Thienen JV, van der Veldt AA, Westgeest HM, Zeijdner EE, Aben KK, van den Hurk C, Zondervan PJ, Bins AD. The PRO-RCC study: a long-term PROspective Renal Cell Carcinoma cohort in the Netherlands, providing an infrastructure for 'Trial within Cohorts' study designs. BMC Cancer. 2023 Jul 11;23(1):648. doi: 10.1186/s12885-023-11094-9. PMID 37434119
- See also: official study and foundation website — http://www.pro-rcc.nl